CLINICAL TRIAL: NCT00896285
Title: TIME1: A 2 X 2 Factorial Trial to Assess Whether Non-steroidal Anti-inflammatory Analgesics and Small-bore Chest Tubes Are Less Painful Than Opiate Analgesics and Large-bore Chest Tubes in Pleurodesis for Malignant Pleural Effusion.
Brief Title: The First Therapeutic Intervention in Malignant Pleural Effusion Trial
Acronym: TIME-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 200816478
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2015-07-20 (Estimated); Status verified 2015-07

CONDITIONS: Malignant Pleural Effusion; Pleural Effusion
Keywords: Pleural malignancy; pleural effusion; pleurodesis; chest tube; cancer; cancer pain management
MeSH Terms: conditions — Pleural Effusion, Malignant; Pleural Effusion; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator)
  Interventions: Other: Large bore chest drain + NSAID based analgesic regimen
- 2 (Active Comparator)
  Interventions: Other: Small bore chest drain + NSAID based analgesic regimen
- 3 (Active Comparator)
  Interventions: Other: Large bore chest drain + opiate based analgesic regimen
- 4 (Active Comparator)
  Interventions: Other: Small bore chest drain + opiate based analgesic regimen

INTERVENTIONS:
Other: Large bore chest drain + NSAID based analgesic regimen — Chest tube greater than 14 French size and ibuprofen.
  Arms: 1
Other: Small bore chest drain + NSAID based analgesic regimen — Chest tube less than or equal to 14 French size and ibuprofen.
  Arms: 2
Other: Large bore chest drain + opiate based analgesic regimen — Chest tube greater than 14 French size and morphine.
  Arms: 3
Other: Small bore chest drain + opiate based analgesic regimen — Chest tube less than or equal to 14 French size and morphine.
  Arms: 4

SUMMARY:
Fluid caused by cancer cells may accumulate in the lining of the lung. Draining the fluid with a chest tube may relieve pain and shortness of breath. To stop the fluid from coming back again, patients are given a medicine (talc) into the chest drain to seal up the space around the lung. This procedure is known as pleurodesis. This sometimes causes pain and discomfort, and the investigators do not know the best way of preventing this.

The investigators hope to find the best way to prevent pain during pleurodesis.

DETAILED DESCRIPTION:
Patients with metastatic cancer often have fluid collecting around the lung as a result of cancer cells spreading to the membranes adjacent to the lung (malignant pleural effusion). The standard way of treating this condition, which may cause unpleasant symptoms such as breathlessness and cough, is to drain the fluid off and then seal the cavity, using a drug (talc) given into the chest drain. Talc causes inflammation in the lining of the lung and chest wall, sticking the two surfaces together and preventing fluid from recurring. This procedure is often very painful; the pain may be partly related to the size of the chest tube used and the type of analgesia taken by the patient during the procedure. Reducing the amount of pain associated with this procedure would be a substantial benefit for patients undergoing this procedure.

This trial is looking at which of two different drug regimens is more effective in preventing pleurodesis pain, and whether the size of chest tube influences pain. It will also address whether either of these influences success rate of pleurodesis.

We hope to learn whether the size of chest drain or the type of pain medication given (ibuprofen or morphine) influences the amount of pain felt after the pleurodesis procedure. We hope to find the best way of preventing pain during this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically confident diagnosis of malignant pleural effusion requiring pleurodesis. The diagnosis may be established by one of:

   * Histologically proven pleural malignancy OR
   * Typical features of pleural malignancy seen on direct vision during thoracoscopy OR
   * Pleural effusion in the context of histologically proven cancer elsewhere
2. Expected survival more than 1 month
3. Written informed consent

Exclusion Criteria:

1. Age < 18 years
2. Primary lymphoma or small cell lung carcinoma
3. Patients who are pregnant or lactating
4. Inability to give informed consent
5. History of GI bleeding or of untreated peptic ulceration
6. Known sensitivity to non-steroidal anti-inflammatory drugs (NSAIDs)/opiates/acetaminophen
7. Hypercapnic respiratory failure
8. Known intravenous drug abuse
9. Severe renal or liver disease
10. Known bleeding diathesis
11. Warfarin therapy
12. Current or recent (within 2 weeks) corticosteroid steroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
An average pain score over 72 hours post pleurodesis for malignant pleural effusion | 72 hours
Pleurodesis success at 3 months post randomization (time to relapse of pleural effusion) | 3 months

SECONDARY OUTCOMES:
Presence of chronic chest pain on the side of the pleurodesis | 6 weeks
Presence of chronic chest pain on the side of the pleurodesis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: RJO Davies, Dr., Principal Investigator — Oxford Pleural Unit, Churchill Hospital, Oxford, England
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States